CLINICAL TRIAL: NCT01490359
Title: South African Men Health Promotion Project
Brief Title: Men Together Making a Difference: Reducing HIV/STD Risk Behavior Among South African Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Fort Hare (Other); Temple University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, John Jemmott, Kenneth B. Clark Professor of Communication in Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 806038; 1R01HD053270 (NIH)
Record Dates: First submitted 2011-12-07; First posted 2011-12-13 (Estimated); Results first posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Human Immunodeficiency Virus Infection; Sexually Transmitted Diseases
Keywords: human immunodeficiency virus; randomized controlled trial; intervention studies; South Africa; men; sexually behavior; social cognitive theory
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were masked to intervention arm at time of recruitment.
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV/STD risk-reduction (Experimental): Men Making a Difference HIV/STD Risk Reduction Intervention was designed to reduce sexual risk behaviors that increase risk of HIV and other sexually transmitted diseases.
  Interventions: Behavioral: Men Making a Difference HIV/STD Risk Reduction Intervention
- Health Promotion Control (Active Comparator): Health Promotion Intervention was designed to increase physical activity, healthful diet, and other behaviors to reduce risk of noncommunicable diseases, including diabetes, hypertension, and cancers.
  Interventions: Behavioral: Health Promotion Control

INTERVENTIONS:
Behavioral: Men Making a Difference HIV/STD Risk Reduction Intervention — Developed based on social cognitive theory and extensive formative research, Men Together Making a Difference HIV/STD risk-reduction intervention consists of 6 75-minute modules designed to increase beliefs that support condom use; skill and self-efficacy to use condoms; and HIV/STD risk-reduction knowledge. Two modules are implemented in each of 3 weekly sessions. It is highly structured and implemented in small groups of 9 to 15 men led by a male, isiXhosa-speaking facilitators using standardized intervention manuals. It includes interactive exercises, games, brainstorming, role-playing, take-home assignments, group discussions, and videos, produced specifically for the interventions, shot in authentic township settings, including a shebeen (i.e., an informal alcohol outlet).
  Other Names: HIV/STD Risk Reduction Intervention
  Arms: HIV/STD risk-reduction
Behavioral: Health Promotion Control — The health-promotion intervention was designed to control for non-specific features including group interaction and special attention. It was structurally similar to the HIV/STD risk-reduction intervention in that it contained activities similar to the HIV/STD risk-reduction intervention but focused on behaviors linked to the risk of heart disease, hypertension, stroke, diabetes, and certain cancers-leading causes of morbidity and mortality among South Africans. It also consisted of 6 75-minute modules implemented 2 modules per week during 3 weekly sessions led by isiXhosa speaking male facilitators. It was designed to increase fruit and vegetable consumption and physical activity and decrease excessive alcohol consumption.
  Other Names: Attention-Control
  Arms: Health Promotion Control

SUMMARY:
Sub-Saharan Africa has about 10% of the world's population, but was home to more than 60% of all people living with HIV in 2003. South Africa continues to have the largest number of people living with HIV in the world, and as in other parts of sub-Saharan Africa, heterosexual exposure is the primary HIV transmission category. Worldwide, efforts to stem the spread of HIV among heterosexuals have stressed the impact of HIV on women. Oft-cited statistics indicate that about half of all people living with HIV are women. The strategies typically offered to address the impact of HIV on women are interventions with women. An alternative approach to addressing women's risk of heterosexual transmission of HIV, one that would be an important complement to the predominant approach, is focusing on men. By reducing sexual risk behavior of men, it should be possible to reduce rates of HIV in both men and women. The rates in men would decline because they are the recipients of the intervention; rates in women would decline because they have sex with men. Interventions aimed at men could take into account the power that men have in sexual decision-making and risk taking. However, whether one considers the US literature or the international literature, few randomized controlled trials of HIV/STD risk-reduction interventions have focused on heterosexual men. Accordingly, the purpose of this research is to develop and test the efficacy of an intervention to curb HIV/STD risk-associated behavior in South African men who have sex with women. A cluster-randomized controlled trial design will be used to reduce the potential for contamination between treatment arms that would be present if individuals were randomized. An attention control group will be used to control for Hawthorne effects, special attention, and group interaction. Matched pairs of neighborhoods in Black townships in Eastern Cape Province, South Africa similar on key characteristics will be created, 22 pairs will be randomly selected, and men will be recruited. One neighborhood in each pair will be randomly assigned to each of the 2 study arms. We hypothesized that men who receive a culturally appropriate theory-based HIV/STD risk-reduction intervention will be more likely to report consistently using condoms during intercourse in the 12-month post intervention period than will men who receive an attention-control intervention, adjusting for baseline condom use.

DETAILED DESCRIPTION:
Sub-Saharan Africa has just over 10% of the world's population, but according to UNAIDS was home to more than 60% of all people living with HIV in 2003-some 25.4 million people. South Africa continues to have the largest number of people living with HIV in the world. As in other parts of sub-Saharan Africa, heterosexual exposure is the primary HIV transmission category. An estimated 5.3 million South Africans-2.9 million women and 2.4 million men-were living with HIV at the end of 2003.

Worldwide, efforts to stem the spread of HIV among heterosexuals have stressed the impact of HIV on women. Oft-cited statistics indicate that about half of all people living with HIV are women. It is often suggested that women are seldom free to make empowered choices and face a range of HIV-related vulnerabilities that men do not face-many of which are embedded in the social relations and economic realities of their societies. Women's economic dependence on their male partners and the fact that women do not have the power to abstain from sex or to insist on condom use-even when they suspect that their man has other sexual partners and might have HIV-is emphasized. The hazards of young women's sexual relationships with older men and the high rate of rape and other forms of sexual coercion are cited. Men are typically mentioned as injection drug users, as having sex with other men-whether as MSMs or being on the "down low"-or as being the cause of the spread of HIV in women. The strategies typically offered to address the impact of HIV on women are interventions with women. For instance, it is recommended that women be taught the information and skills to make decisions about the terms of their sexual relationships, that methods of protection that women can control (e.g., microbicides) be developed, and that boosting women's economic opportunities and social power should be seen as part and parcel of potentially successful and sustainable HIV prevention strategies.

To be sure, there is an alternative approach to addressing women's risk of heterosexual transmission of HIV, one that would be important complement to the predominant approach: namely, focusing on men. Although it is noted that HIV is affecting women most severely in places where heterosexual exposure is a dominant mode of transmission, this seldom leads to a recommendation that interventions be developed to change men's behavior. Yet, by reducing men's sexual risk behavior, it should be possible to reduce rates of HIV in both men and women. Men's rates would decline because they are the recipients of the intervention; women's rates would decline because they have sex with men. Interventions targeting men could take into account the power that men have in sexual decision-making and risk taking.

However, whether one considers the US literature or the international literature, few randomized controlled trials (RCTs) of HIV/STD risk-reduction interventions have targeted heterosexual men. Elwy and colleagues 2002 review of HIV/STD prevention intervention studies revealed that only 12 of 1157 studies worldwide were conducted on males only. Most were not RCTs demonstrating intervention efficacy. Only 2 demonstrated significant effects on mediators and behaviors, and neither was a RCT. In addition, scant attention has focused on the general population of heterosexual men in any region. Indeed, 8 of the 12 studies focused on incarcerated men, STD patients, substance abusers, miners, or truck drivers. To address this gap in the literature, the proposed trial will focus on men who are more representative of the general population. In many developing countries, including South Africa, the HIV/AIDS epidemic is generalized, and there is a need to develop and test interventions for a broad range of the population, not just special high-risk sub-populations.

Accordingly, the purpose of this research is to develop and test the efficacy of an intervention to reduce behaviors that create the risk for contracting and transmitting STD, including HIV, among South African men who have sex with women. A cluster-randomized control trial design will be used to reduce the potential for contamination between treatment arms that would be present if individuals were randomized. An attention control group will be used to control for Hawthorne effects, special attention, and group interaction. Men will be recruited from Black townships surrounding East London, including Mdantsane, Scenery Park, Duncan, Village, and Gompo Town, and the semi-rural area of Berlin in the Eastern Cape Province of South Africa. More than 98% of the residents of these areas are Black Africans, and isiXhosa is the first language for 98.8% of the population. There are 206 neighborhoods defined as geographical clusters tied to census data in this catchment area, allowing the creation of 103 matched pairs of neighborhoods similar on the percentage isiXhosa-speaking, percentage married, percentage male, percentage living in informal dwellings, percentage unemployed, and population size. From the 103 matched pairs, 22 pairs will be randomly selected for the trial. One neighborhood in each pair will be randomly assigned to each of the 2 study arms.

Before recruiting from a neighborhood, meetings with community leaders (e.g., councilor, clergy) will be held to enlist their support. In addition, a meeting will be held to inform men in the neighborhood about the study. Recruiters will inform potential participants about the study, obtain consent to be screened, and conduct a brief screening interview to determine eligibility and willingness to participate. Eligible men will be invited to participate in the "Men, Together Making A Difference Project" designed to understand men's behaviors that may create health risks such as heart disease, cancer, and STDs, especially HIV, and to find ways to teach men how to reduce these risks. A common participant recruitment and enrollment protocol, including use of the same posters and other materials, will be followed in the neighborhoods in both conditions. Eligible men will be recruited in advance of randomization so that at the time they agree to participate they will be blind to the specific intervention they will receive. This procedure will reduce the probability of self-selection bias into the different conditions of the trial.

All participants will complete self-report measures via audio computer-assisted self-interviewing before the intervention, immediately after, and 6 and 12 months after the intervention. Several steps will be taken to increase the validity of self-report measures. Participants will be given a calendar, with the dates clearly marked. This will make salient to respondents the dates that are included when they are asked to recall their behavior "in the past 3 months" and that they should be specific. The importance of responding honestly will be emphasized. They will be informed that their responses will be used to create programs for South African men like themselves and that this will be possible only if they answer the questions honestly. This pits the social responsibility motive against the social desirability motive. Participants will be assured that their responses will be kept confidential. Facilitators who lead the intervention groups will not be involved in any way in the data collection. The use of ACASI should also serve to increase participants' motivation to respond accurately.

There are 2 Specific Aims. Aim 1 is to test the primary hypothesis that men who receive a culturally appropriate theory-based HIV/STD risk-reduction intervention will be more likely to report consistently using condoms during vaginal intercourse in the 12-month post intervention period than will men who receive an attention-control intervention. Aim 2 is to test the secondary hypothesis that outcome expectancies and self-efficacy to use condoms mediate the HIV/STD risk-reduction intervention's effect on condom use. In addition, an exploratory aim is to conduct hypothesis-generating analyses on whether the efficacy of the intervention varies depending on neighborhood characteristics or participants' baseline characteristics. The effects of HIV/STD risk-reduction interventions may differ as a function of the neighborhood's unemployment rate, percentage living in informal dwellings/shacks, percentage married, or sex ratio. Potential individual-level moderators include age, marital status, language use (English versus isiXhosa), and alcohol and drug use.

The unit of inference in this trial is the individual. This is because the trial is designed to test the efficacy of a behavior-change intervention based on individual-level behavior change theory. As Donner and Klar in 2000 noted in their influential textbook on cluster-randomized trial, the unit of inference, not the unit of randomization, determines the unit of analysis.

The data will be analyzed using an intention-to-treat mode, with participants analyzed based on their intervention assignment, regardless of the number of intervention or data-collection sessions attended. The primary aim focuses on testing for significant differences between two treatment conditions over the post intervention period. Major statistical challenges arise in the proper handling of repeated clustered outcomes. Each variable of interest is completed by each man, nested within a neighborhood, thus creating a correlated outcome. Moreover, the multiple assessments of each variable over the study period produce correlated repeated outcomes. The primary challenge in the analysis of such data is appropriate adjustments for the differential treatment means between clusters and the correlations among the observations within a cluster (cluster effects).

Most statistical models assume stochastic independence among observations and thus are inappropriate for clustered data. In this trial, generalized estimating equations (GEE) modeling will be employed to handle the clustered data appropriately. GEE modeling avoids explicit modeling of the within-cluster correlations by basing statistical inferences of model parameters on marginalized likelihood or generalized estimating equations. Since GEE requires a relatively large sample size, it is not appropriate for small studies. Given the large sample size, GEE is appropriate for in this trial. The implementation for this trial is relatively straightforward. For instance, to determine whether a greater percentage of the men who receive the HIV/STD risk-reduction intervention report consistent condom use 6 and 12 months post intervention, as compared with those who received the health-promotion intervention, the model will include time-independent covariates, baseline measure of consistent condom use, intervention type, and time (2 categories representing 6- and 12-month follow-up), which will provide the effect of the intervention over the 2 follow-up visits.

A sample size calculation was performed to detect an a priori effect size of a 10% increase in consistent condom use from 32% to 42% in the HIV/STD risk-reduction intervention condition, adjusting for the expected variance inflation due to clustering. A 10% increase was selected as a clinically and substantively important effect size. Based on pilot data, an intraclass correlation (ICC) of 0.01 was estimated. Assuming alpha = 0.05, a 2-tailed test, ICC = 0.01, 15% attrition at 12-month follow-up, and N = 1,152 men in the trial from 44 neighborhoods with an average of 26 men in each neighborhood, the trial was estimated to have 81% power to detect a 10% increase in consistent condom use from 32% to 42% in the HIV/STD intervention group. Assuming the same effect size, hypothesis tests on secondary sexual behavior outcomes and theoretical mediator variables will have similar statistical power.

ELIGIBILITY:
Inclusion Criteria:

* Men ages 18 to 45 years
* Reside in a randomly selected neighborhoods
* Report vaginal intercourse in the previous 3 months
* Have a photo identification

Exclusion Criteria:

* Plan to relocate from the area within the next 15 months

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1181 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John B Jemmott III, PhD, Principal Investigator — Trustees of the University of Pennsylvania

REFERENCES:
- [Background] Icard LD, Jemmott JB 3rd, Teitelman A, O'Leary A, Heeren GA. Mediation effects of problem drinking and marijuana use on HIV sexual risk behaviors among childhood sexually abused South African heterosexual men. Child Abuse Negl. 2014 Feb;38(2):234-42. doi: 10.1016/j.chiabu.2013.08.002. Epub 2013 Sep 13. PMID 24041455
- [Background] Heeren GA, Icard LD, O'Leary A, Jemmott JB 3rd, Ngwane Z, Mtose X. Protective factors and HIV risk behavior among South African men. AIDS Behav. 2014 Oct;18(10):1991-7. doi: 10.1007/s10461-014-0767-2. PMID 24722765
- [Result] Jemmott JB 3rd, Jemmott LS, O'Leary A, Ngwane Z, Icard LD, Heeren GA, Mtose X, Carty C. Cluster-randomized controlled trial of an HIV/sexually transmitted infection risk-reduction intervention for South African men. Am J Public Health. 2014 Mar;104(3):467-73. doi: 10.2105/AJPH.2013.301578. Epub 2014 Jan 16. PMID 24432923
- [Result] O'Leary A, Jemmott JB 3rd, Jemmott LS, Bellamy S, Icard LD, Ngwane Z. Mediation of an efficacious HIV risk reduction intervention for South African men. AIDS Behav. 2015 Oct;19(10):1842-9. doi: 10.1007/s10461-015-1042-x. PMID 25969177
- [Result] Jemmott JB 3rd, Jemmott LS, Ngwane Z, Zhang J, Heeren GA, Icard LD, O'Leary A, Mtose X, Teitelman A, Carty C. Theory-based behavioral intervention increases self-reported physical activity in South African men: a cluster-randomized controlled trial. Prev Med. 2014 Jul;64:114-20. doi: 10.1016/j.ypmed.2014.04.012. Epub 2014 Apr 13. PMID 24736094
- [Result] Jemmott JB 3rd, Stephens-Shields A, O'Leary A, Jemmott LS, Teitelman A, Ngwane Z, Mtose X. Mediation of effects of a theory-based behavioral intervention on self-reported physical activity in South African men. Prev Med. 2015 Mar;72:1-7. doi: 10.1016/j.ypmed.2014.12.022. Epub 2015 Jan 4. PMID 25565482

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV/STD Risk-reduction: Men Making a Difference HIV/STD Risk Reduction Intervention was designed to reduce sexual risk behaviors that increase risk of HIV and other sexually transmitted diseases.
  Men Making a Difference HIV/STD Risk Reduction Intervention: Developed based on social cognitive theory and extensive formative research, it consists of 6 75-minute modules designed to increase beliefs that support condom use; skill and self-efficacy to use condoms; and HIV/STD risk-reduction knowledge. Two modules are implemented in each of 3 weekly sessions. It is highly structured and implemented in small groups of 9 to 15 men led by a male, isiXhosa-speaking facilitators using standardized intervention manuals. It includes interactive exercises, games, brainstorming, role-playing, take-home assignments, group discussions, and videos, produced specifically for the interventions, shot in authentic township settings, including a shebeen (i.e., an informal alcohol outlet).
Period: Overall Study
Arm/Group | HIV/STD Risk-reduction | Health Promotion Control
Started | 609 | 572
Followed-up at 6 mo | 558 | 535
Followed-up at 12 mo | 569 | 537
Completed | 585 | 555
Not Completed | 24 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV/STD Risk-reduction | Health Promotion Control | Total
Number analyzed (Participants) | 609 | 572 | 1181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 609 | 572 | 1181
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 609 | 572 | 1181
Race/Ethnicity, Customized [Number; unit: participants]
  Black South African | 609 | 572 | 1181
  Not Black South African | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 609 | 572 | 1181
Married [Number; unit: participants]
  Married | 27 | 41 | 68
  Not Married | 582 | 531 | 1113
Employment Status [Number; unit: participants]
  Not employed | 425 | 368 | 793
  Employed | 184 | 204 | 388
Completed high school [Number; unit: participants]
  Completed high school | 279 | 239 | 518
  Less than high school | 330 | 333 | 663
Alcohol dependent [Number; unit: participants]
  Alcohol dependent | 377 | 330 | 707
  Not alcohol dependent | 232 | 242 | 474

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Consistent Condom Use During Vaginal Intercourse in the Past 3 Months
Description: Men who reported at least 1 vaginal intercourse act in the past 3 months and whose number of reported condom-protected vaginal intercourse acts equaled their number of vaginal intercourse acts were coded as practicing consistent or 100% condom use. Men who reported at least 1 vaginal intercourse act and whose reported number of condom-protected vaginal intercourse acts was less than their number of vaginal intercourse acts were coded as not practicing consistent condom use. Separate binary variables reflected consistent condom use with primary partners and casual partners.
Time Frame: Baseline, 6 months, 12 months post-intervention
Population: Participants with data at baseline and at least one follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV/STD Risk-reduction | Health Promotion Control
Number analyzed (Participants) | 418 | 387
Participants
  Baseline steady partner: number analyzed (Participants) | 365 | 325
  Baseline steady partner | 121 | 103
  6 mo steady partner: number analyzed (Participants) | 311 | 273
  6 mo steady partner | 125 | 93
  12 mo steady partner: number analyzed (Participants) | 299 | 274
  12 mo steady partner | 119 | 81
  Baseline casual partners: number analyzed (Participants) | 151 | 142
  Baseline casual partners | 91 | 78
  6 mo casual partners: number analyzed (Participants) | 109 | 104
  6 mo casual partners | 60 | 58
  12 mo casual partners: number analyzed (Participants) | 104 | 96
  12 mo casual partners | 56 | 48
Statistical Analysis 1: Comparison: HIV/STD Risk-reduction vs Health Promotion Control; Assuming alpha = 0.05, a 2-tailed test, ICC = 0.01, 15% attrition at 12-month follow-up, and N = 1,152 men in the trial from 44 neighborhoods with an average of 26 men in each neighborhood, the trial was estimated to have 81% power to detect a 10% increase in consistent condom use from 32% to 42% in the HIV/STI intervention group; Test type: Superiority or Other; p = .008, generalized estimating equations (GEE) — The GEE model included baseline measure of consistent condom use, intervention condition, time (6- vs. 12-mo follow-up), and type of partner (steady vs casual partners) with robust standard errors and an independent working correlation matrix; Odds Ratio (OR) = 1.32, 95% CI 2-sided [1.03 to 1.71] — Estimate is odds ratio (intervention vs. health control)

2. Secondary Outcome: The Self-reported Proportion of Condom-protected Acts of Vaginal Intercourse in the Past 3 Months
Description: The proportion of condom-protected acts of vaginal intercourse is defined as the self-reported number of acts of vaginal intercourse in which the respondent used a condom in the past 3 months divided by the total number of acts of vaginal intercourse the respondent reported in the past 3 months. Calculated separately for steady and casual partners.
Time Frame: Baseline, 6 months, 12 months post intervention
Population: Participants with data at baseline and at least one post-intervention assessment.
Measure: Mean (Standard Error); unit: proportion of acts
Groups:
- HIV/STD Risk-reduction: Men Making a Difference HIV/STD Risk Reduction Intervention was designed to reduce sexual risk behaviors that increase risk of HIV and other sexually transmitted diseases.
  Men Making a Difference HIV/STD Risk Reduction Intervention: Developed based on social cognitive theory and extensive formative research, the intervention consists of 6 75-minute modules designed to increase beliefs that support condom use; skill and self-efficacy to use condoms; and HIV/STD risk-reduction knowledge. Two modules are implemented in each of 3 weekly sessions. It is highly structured and implemented in small groups of 9 to 15 men led by a male, isiXhosa-speaking facilitators using standardized intervention manuals. It includes interactive exercises, games, brainstorming, role-playing, take-home assignments, group discussions, and videos, produced specifically for the interventions, shot in authentic township settings, including a shebeen (i.e., an informal alcohol outlet).
Arm/Group | HIV/STD Risk-reduction | Health Promotion Control
Number analyzed (Participants) | 418 | 387
proportion of acts
  Baseline Steady partners: number analyzed (Participants) | 365 | 325
  Baseline Steady partners | 0.524 (0.021) | 0.516 (0.022)
  Baseline Casual partners: number analyzed (Participants) | 151 | 142
  Baseline Casual partners | 0.713 (0.024) | 0.665 (0.028)
  6 mo Steady partners: number analyzed (Participants) | 311 | 273
  6 mo Steady partners | 0.585 (0.022) | 0.549 (0.023)
  6 mo Casual partners: number analyzed (Participants) | 109 | 104
  6 mo Casual partners | 0.712 (0.029) | 0.685 (0.029)
  12 mo Steady partners: number analyzed (Participants) | 299 | 274
  12 mo Steady partners | 0.613 (0.021) | 0.555 (0.022)
  12 mo Casual partners: number analyzed (Participants) | 104 | 96
  12 mo Casual partners | 0.678 (0.031) | 0.684 (0.030)

3. Secondary Outcome: Self-reported Condom Use at Most Recent Vaginal Intercourse
Description: The respondents' self-report of using a condom during their most recent vaginal intercourse. Calculated separately for steady and casual partners.
Time Frame: Baseline, 6 months, 12 months post intervention
Population: Participants with data at baseline and at least one post-intervention assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV/STD Risk-reduction | Health Promotion Control
Number analyzed (Participants) | 418 | 387
Participants
  Baseline Steady partners: number analyzed (Participants) | 365 | 325
  Baseline Steady partners | 193 | 175
  Baseline Casual partners: number analyzed (Participants) | 151 | 143
  Baseline Casual partners | 119 | 108
  6 mo Steady partners: number analyzed (Participants) | 311 | 273
  6 mo Steady partners | 216 | 162
  6 mo Casual partners: number analyzed (Participants) | 109 | 105
  6 mo Casual partners | 96 | 85
  12 mo Steady partners: number analyzed (Participants) | 299 | 274
  12 mo Steady partners | 204 | 176
  12 mo Casual partners: number analyzed (Participants) | 104 | 96
  12 mo Casual partners | 80 | 75

4. Secondary Outcome: Frequency of Condom Use in the Past 3 Months
Description: Respondents' rating on a 5-point scale from 1 (never) to 5 (always) how often they used a condom during vaginal intercourse. Measured separately for steady and casual partners.
Time Frame: Baseline, 6 months, 12 months post intervention
Population: Participants with data from baseline and at least one post-intervention assessment.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | HIV/STD Risk-reduction | Health Promotion Control
Number analyzed (Participants) | 418 | 387
units on a scale
  Baseline Steady partners: number analyzed (Participants) | 365 | 325
  Baseline Steady partners | 2.991 (0.078) | 3.041 (0.083)
  Baseline Casual partners: number analyzed (Participants) | 151 | 142
  Baseline Casual partners | 3.712 (0.093) | 3.603 (0.109)
  6 mo Steady partners: number analyzed (Participants) | 311 | 273
  6 mo Steady partners | 3.309 (0.079) | 2.931 (0.085)
  6 mo Casual partners: number analyzed (Participants) | 109 | 104
  6 mo Casual partners | 3.892 (0.101) | 3.594 (0.110)
  12 mo Steady partners | 3.238 (0.077) | 3.029 (0.081)
  12 mo Casual partners: number analyzed (Participants) | 104 | 96
  12 mo Casual partners | 3.702 (0.109) | 3.649 (0.111)

5. Secondary Outcome: Talked to Partner About Condom Use
Description: A binary variable indicating whether the participants talked to partner about using condoms in the past 90 days.
Time Frame: Baseline, 6 months, 12 months post intervention
Population: Participants with data at baseline and at least one post-intervention assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV/STD Risk-reduction | Health Promotion Control
Number analyzed (Participants) | 490 | 466
Participants
  Baseline Steady partners: number analyzed (Participants) | 425 | 390
  Baseline Steady partners | 318 | 269
  Baseline Casual partners: number analyzed (Participants) | 220 | 192
  Baseline Casual partners | 145 | 124
  6 mo Steady partners: number analyzed (Participants) | 369 | 329
  6 mo Steady partners | 310 | 243
  6 mo Casual partners: number analyzed (Participants) | 163 | 149
  6 mo Casual partners | 122 | 100
  12 mo Steady partners: number analyzed (Participants) | 360 | 335
  12 mo Steady partners | 294 | 245
  12 mo Casual partners: number analyzed (Participants) | 150 | 130
  12 mo Casual partners | 105 | 90

6. Secondary Outcome: Condomless Vaginal Intercourse in the Past 3 Months
Description: A binary variable indicating whether participant reported having vaginal intercourse without using a condom in the past 3 months (0 = did not have vaginal intercourse or always used a condom; 1= did have vaginal intercourse without using a condom)
Time Frame: Baseline, 6 months, and 12 months post-intervention
Population: Participants with data at baseline and at least one post-intervention assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV/STD Risk-reduction | Health Promotion Control
Number analyzed (Participants) | 585 | 555
Participants
  Baseline steady partner | 281 | 263
  6 mo steady partner: number analyzed (Participants) | 558 | 535
  6 mo steady partner | 231 | 220
  12 mo steady partner: number analyzed (Participants) | 566 | 537
  12 mo steady partner | 231 | 230
  Baseline casual partner: number analyzed (Participants) | 585 | 554
  Baseline casual partner | 112 | 107
  6 mo casual partner: number analyzed (Participants) | 558 | 534
  6 mo casual partner | 82 | 83
  12 mo casual partner: number analyzed (Participants) | 567 | 535
  12 mo casual partner | 84 | 83

7. Secondary Outcome: Heterosexual Anal Intercourse in the Past 3 Months
Description: The report of having anal intercourse with a woman in the past 3 months
Time Frame: Baseline, 6 months, 12 months post intervention
Population: Participants with data at baseline and at least one post-intervention assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV/STD Risk-reduction | Health Promotion Control
Number analyzed (Participants) | 568 | 543
Participants
  Baseline Steady partners: number analyzed (Participants) | 547 | 527
  Baseline Steady partners | 59 | 58
  Baseline Casual partners: number analyzed (Participants) | 517 | 482
  Baseline Casual partners | 41 | 35
  6 mo Steady partners: number analyzed (Participants) | 512 | 493
  6 mo Steady partners | 42 | 48
  6 mo Casual partners: number analyzed (Participants) | 463 | 444
  6 mo Casual partners | 25 | 31
  12 mo Steady partners: number analyzed (Participants) | 520 | 503
  12 mo Steady partners | 35 | 35
  12 mo Casual partners: number analyzed (Participants) | 484 | 453
  12 mo Casual partners | 20 | 18

8. Secondary Outcome: Multiple Vaginal Partners in the Past 3 Months
Description: The report of having vaginal intercourse with 2 or more women in the past 3 months.
Time Frame: Baseline, 6 months, 12 months post intervention
Population: Participants with data at baseline and at least one post-intervention assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV/STD Risk-reduction | Health Promotion Control
Number analyzed (Participants) | 585 | 554
Participants
  Baseline | 256 | 220
  6 mo: number analyzed (Participants) | 558 | 534
  6 mo | 199 | 191
  12 mo: number analyzed (Participants) | 567 | 536
  12 mo | 199 | 200

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | HIV/STD Risk-reduction | Health Promotion Control
Serious Adverse Events (participants affected / at risk) | 0/609 | 0/572
Other Adverse Events (participants affected / at risk) | 0/609 | 0/572

LIMITATIONS AND CAVEATS:
A limitation of the study is the reliance on self-reports of behavior. In addition, the results may not generalize to all South African men.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes